CLINICAL TRIAL: NCT01899534
Title: Mental Health E-screening in Pregnant and Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dawn Kingston, Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00039130
Record Dates: First submitted 2013-07-10; First posted 2013-07-15 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Depression; Anxiety
Keywords: Pregnancy; Mental Health; Screening; Computer; Feasibility
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paper-based screening (No Intervention): Paper-based screening. Women will complete a mental health screening tool on paper (usual care).
- E-screening (Experimental): Women will complete mental health screening on a tablet
  Interventions: Other: E-screening

INTERVENTIONS:
Other: E-screening — E-screening will be conducted on a computer tablet with wireless access. The tablet will be configured with the screening tool currently used in each clinic. The content and order of individual questions will be identical to the paper-pen version. Response options will be listed in full view under each question. Women select responses by touching the screen.
  Arms: E-screening

SUMMARY:
To compare e-screening versus usual screening on: 1) women's and healthcare providers' views on feasibility and acceptability; 2) rates of detection of prenatal and postpartum depression and anxiety; 3) perceived risk and benefit of disclosure; 4) cost-effectiveness; 5) psychometric properties. We also aim to identify factors associated with feasibility of e-screening.Compared to usual screening:1) e-screening is as feasible; 2) e-screening yields similar rates of prenatal and postpartum depression and anxiety; 3) the mean score for risk of disclosure is significantly lower and benefit of disclosure is significantly higher in the e-screening group; 4) e-screening is as or more cost effective in detecting prenatal and postpartum depression and anxiety; 5) features of e-screening are significantly associated with feasibility and acceptability, whereas demographic factors are not; and 6) reliability and validity indices of ALPHA and EPDS are strongly correlated for both administration modes.

DETAILED DESCRIPTION:
Given that it is critical to conduct screening within a system that links referral and treatment, our IMPACT pilot trial is evaluating integrated screening and care (see Summary of Progress) versus usual prenatal care. The proposed trial engages 2 unique clinics with experienced staff who conduct routine screening (with referrals and treatment in place) to evaluate different modalities of screening. Since widespread screening is unlikely to be successfully implemented if it entails additional human resources, this trial assesses the potential for a sustainable, e-health alternative.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and postpartum women will be eligible for this study if they:

  1. receive care at the recruitment sites ;
  2. can read/write English; and
  3. are willing to complete e-screening

Exclusion Criteria:

1. do not receive care at the recruitment site;
2. cannot read/write English;
3. are not willing to complete e-screening

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome is feasibility/acceptability of the process of e-screening (vs 'usual' screening). | 10 months
  All women will complete: 1) the Computer Violence Assessment Evaluation (CVAE) 38 (originally designed The primary outcome is feasibility/acceptability of the process of e-screening (vs 'usual' screening).to evaluate the feasibility/acceptability aspects of e- screening of domestic violence -Appendix C); and 2) open-ended investigator-developed questions on e-screening feasibility currently being pre-tested in another study (Appendix D).

SECONDARY OUTCOMES:
Proportion of pregnant and postpartum women with clinical depression and anxiety. | on recruitment
  Measured in in pregnant women using the Antenatal Psychosocial Health Assessment (ALPHA)and the Edinburgh Postnatal Depression Scale. Measured in pregnant women using the Edinburgh Postnatal Depression Scale.
  self-reported
Depression and anxiety | Within one week of recruitment
  Mini Diagnostic Interview
  -will be conducted either by telephone or in-person by a member of the research team who is a mental health expert
Cost-effectiveness of e-screening | during recruitment
  We will observe the clinic process for a morning to determine the length of time it takes staff to conduct the both the usual screening process as well as the e-screening process (e.g., distribute tablets, follow-up with women). We will also interview the clinic manager to determine the costs of current screening process (e.g., time to screen, physical resources).

OTHER OUTCOMES:
Mean scores on the Perceived Risk and Perceived Utility subscales of DES | on recruitment
  Disclosure Expectations Scale (DES) Self-reported by women

CONTACTS AND LOCATIONS:
Overall Officials: Dawn A Kingston, Ph.D, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - Dickensfield Primary Care Maternity Clinic, Edmonton, Alberta
  - Royal Alexandra Hospital: Lois Hole Hospital for Women, Edmonton, Alberta
  - Sturgeon Primary Care Maternity Clinic, St. Albert, Alberta

REFERENCES:
- [Derived] Kingston D, Biringer A, Veldhuyzen van Zanten S, Giallo R, McDonald S, MacQueen G, Vermeyden L, Austin MP. Pregnant Women's Perceptions of the Risks and Benefits of Disclosure During Web-Based Mental Health E-Screening Versus Paper-Based Screening: Randomized Controlled Trial. JMIR Ment Health. 2017 Oct 20;4(4):e42. doi: 10.2196/mental.6888. PMID 29054833
- [Derived] Kingston D, Austin MP, Veldhuyzen van Zanten S, Harvalik P, Giallo R, McDonald SD, MacQueen G, Vermeyden L, Lasiuk G, Sword W, Biringer A. Pregnant Women's Views on the Feasibility and Acceptability of Web-Based Mental Health E-Screening Versus Paper-Based Screening: A Randomized Controlled Trial. J Med Internet Res. 2017 Apr 7;19(4):e88. doi: 10.2196/jmir.6866. PMID 28389421
- [Derived] Kingston D, McDonald S, Biringer A, Austin MP, Hegadoren K, McDonald S, Giallo R, Ohinmaa A, Lasiuk G, MacQueen G, Sword W, Lane-Smith M, van Zanten SV. Comparing the feasibility, acceptability, clinical-, and cost-effectiveness of mental health e-screening to paper-based screening on the detection of depression, anxiety, and psychosocial risk in pregnant women: a study protocol of a randomized, parallel-group, superiority trial. Trials. 2014 Jan 2;15:3. doi: 10.1186/1745-6215-15-3. PMID 24383441